CLINICAL TRIAL: NCT06603961
Title: Efficacy of Customized Pressure-Guided Elastic Bandages in Preventing Postoperative Edema and Complications in Coronary Artery Bypass Graft (CABG) Patients: A Comparative Study of Compression Therapy and Standard Post-CABG Care.
Brief Title: Prevention of Edema After Coronary Artery Bypass Graft by Customized Pressure-guided Elastic Bandages
Acronym: PEACCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Ratcharnon Srifa, Ratcharnon Srifa, Cardiothoracic Resident, MD, Sub-Investigator, Cardiothoracic Division, Department of Surgery, Siriraj Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 788/2566(IRB1)
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Limb Edema; Surgical Site Infections; Leg Swelling; Compression Bandages; Coronary Artery Bypass Graft; CABG; Saphenectomy; Saphenous Vein; Delayed Wound Healing; Post Operative Complications; Post Operative Surgical Site Infection
Keywords: compression bandages; compression therapy; customized pressure-guided elastic bandages; CABG; coronary arterial bypass graft
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPG-EB group (Active Comparator): The intervention group received Customized-pressure guided elastic bandage for 4 weeks post-operatively.
  Interventions: Device: CPG-EB group
- Standard group (No Intervention): Standard group is the standard of care in post operative CABG surgery patients. This group used elastic bandage for 24 hours or overnight after surgery.

INTERVENTIONS:
Device: CPG-EB group — Customized-pressure guided elastic bandage group
  Arms: CPG-EB group

SUMMARY:
The study aimed to assess the efficacy of customized pressure-guided elastic bandages (CPG-EB) in preventing postoperative edema and complications in Coronary Artery Bypass Graft (CABG) patients. While compression therapy, like compressive stockings, has benefits in preventing edema, concerns about affordability persist. CPG-EB provides optimal sub-bandage pressure, proven effective in venous leg ulcers. Implementing CPG-EB post-CABG could enhance venous blood flow, reducing complications and improving outcomes. Patients were divided into two groups: one with CPG-EB and the other standard post-CABG care. Data collected at 1, 2, and 6 weeks post-surgery assessed swelling and wound complications. Comparative analysis used standardized criteria.

DETAILED DESCRIPTION:
Inclusion Criteria :

1. All patients scheduled for elective coronary artery bypass grafting (CABG) surgery with saphenous vein harvesting from the leg at Siriraj Hospital.
2. Patients aged 18 years and older undergoing CABG surgery with saphenous vein harvesting from the leg at Siriraj Hospital, who willingly consent to participate in the study.

Exclusion Criteria : *

1. Patients with an Ankle-brachial pressure index (ABI) < 0.8
2. Patients with severe leg swelling (pitting edema of grade 3 or higher) or with pre-existing or post-operative heart failure that remains uncontrolled despite diuretic therapy.
3. Patients with occlusive peripheral arterial disease (PAD) or chronic venous insufficiency (CEAP 2s), characterized by significant venous stasis, leg pain, varicose veins, or lymphadenopathy.

ELIGIBILITY:
Inclusion Criteria:

1. All patients scheduled for elective coronary artery bypass grafting (CABG) surgery with saphenous vein harvesting from the leg at Siriraj Hospital.
2. Patients aged 18 years and older undergoing CABG surgery with saphenous vein harvesting from the leg at Siriraj Hospital, who willingly consent to participate in the study.

Exclusion Criteria:

1. Patients with an Ankle-brachial pressure index (ABI) < 0.8
2. Patients with severe leg swelling (pitting edema of grade 3 or higher) or with pre-existing or post-operative heart failure that remains uncontrolled despite diuretic therapy.
3. Patients with occlusive peripheral arterial disease (PAD) or chronic venous insufficiency (CEAP 2s), characterized by significant venous stasis, leg pain, varicose veins, or lymphadenopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-01-19 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
incidence rate of leg swelling | 1, 2 and 6 weeks after CABG surgery
  Chi-square test
Rate of severity level of swelling | 1, 2 and 6 weeks after CABG surgery
  Chi-square test
differences in leg circumference at various locations between preoperative and postoperative measurements between the two groups. | 1, 2 and 6 weeks after CABG surgery
  Independent sample t-test or Mann-Whitney U test

SECONDARY OUTCOMES:
infection rate | 1, 2 and 6 weeks after CABG surgery
  Chi-square test
rate of delayed wound healing | 1, 2 and 6 weeks after CABG surgery
  Chi-square test
rate of numbness | 1, 2 and 6 weeks after CABG surgery
  Chi-square test

CONTACTS AND LOCATIONS:
Overall Officials: Prompak Nitayavardhana, MD, Study Director — Siriraj Hospital
Locations (2):
- Thailand (2):
  - Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Bangkok Noi
  - Siriraj hospital, Bangkok, Bangkok Noi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wells FC, Newsom SW, Rowlands C. Wound infection in cardiothoracic surgery. Lancet. 1983 May 28;1(8335):1209-10. doi: 10.1016/s0140-6736(83)92479-0. PMID 6134001
- [Background] Utley JR, Thomason ME, Wallace DJ, Mutch DW, Staton L, Brown V, Wilde CM, Bell MS. Preoperative correlates of impaired wound healing after saphenous vein excision. J Thorac Cardiovasc Surg. 1989 Jul;98(1):147-9. PMID 2786980
- [Background] Terada Y, Fukuda S, Tohda E, Kigawa I, Wanibuchi Y, Mitsui T. Venous function and delayed leg swelling following saphenectomy in coronary artery bypass grafting. Jpn J Thorac Cardiovasc Surg. 1999 Nov;47(11):559-62. doi: 10.1007/BF03218062. PMID 10614096
- [Background] Sermsathanasawadi N, Chatjaturapat C, Pianchareonsin R, Puangpunngam N, Wongwanit C, Chinsakchai K, Ruangsetakit C, Mutirangura P. Use of customised pressure-guided elastic bandages to improve efficacy of compression bandaging for venous ulcers. Int Wound J. 2017 Aug;14(4):636-640. doi: 10.1111/iwj.12656. Epub 2016 Aug 9. PMID 27502619
- [Background] Reifsnyder T, Bandyk D, Seabrook G, Kinney E, Towne JB. Wound complications of the in situ saphenous vein bypass technique. J Vasc Surg. 1992 May;15(5):843-8; discussion 848-50. doi: 10.1067/mva.1992.36658. PMID 1578540
- [Background] Rabe E, Partsch H, Morrison N, Meissner MH, Mosti G, Lattimer CR, Carpentier PH, Gaillard S, Junger M, Urbanek T, Hafner J, Patel M, Wu S, Caprini J, Lurie F, Hirsch T. Risks and contraindications of medical compression treatment - A critical reappraisal. An international consensus statement. Phlebology. 2020 Aug;35(7):447-460. doi: 10.1177/0268355520909066. Epub 2020 Mar 2. PMID 32122269
- [Background] Paletta CE, Huang DB, Fiore AC, Swartz MT, Rilloraza FL, Gardner JE. Major leg wound complications after saphenous vein harvest for coronary revascularization. Ann Thorac Surg. 2000 Aug;70(2):492-7. doi: 10.1016/s0003-4975(00)01414-4. PMID 10969669
- [Background] O'Hagan B, Kolvekar S. Use of support stockings after cardiac surgery. Prof Nurse. 2000 Jul;15(10):660-2. PMID 12026465
- [Background] Mountney J, Wilkinson GA. Saphenous neuralgia after coronary artery bypass grafting. Eur J Cardiothorac Surg. 1999 Oct;16(4):440-3. doi: 10.1016/s1010-7940(99)00294-8. PMID 10571092
- [Background] Mosti G, Iabichella ML, Partsch H. Compression therapy in mixed ulcers increases venous output and arterial perfusion. J Vasc Surg. 2012 Jan;55(1):122-8. doi: 10.1016/j.jvs.2011.07.071. Epub 2011 Sep 23. PMID 21944912
- [Background] Mosti G, Cavezzi A. Compression therapy in lymphedema: Between past and recent scientific data. Phlebology. 2019 Sep;34(8):515-522. doi: 10.1177/0268355518824524. Epub 2019 Jan 9. No abstract available. PMID 30626269
- [Background] Lommerud S, Hofoss D. Leg wound infection after coronary artery bypass grafting: A natural experiment comparing use and non-use of a compression stocking. Eur J Cardiovasc Nurs. 2017 Feb;16(2):136-142. doi: 10.1177/1474515116641298. Epub 2016 Jul 8. PMID 27036953
- [Background] Liehr P, Todd B, Rossi M, Culligan M. Effect of venous support on edema and leg pain in patients after coronary artery bypass graft surgery. Heart Lung. 1992 Jan;21(1):6-11. PMID 1735659
- [Background] Khoshgoftar Z, Ayat Esfahani F, Marzban M, Salehi Omran A, Haji Ghasemi A, Movaghar S, Saadat S. Comparison of compression stocking with elastic bandage in reducing postoperative edema in coronary artery bypass graft patient. J Vasc Nurs. 2009 Dec;27(4):103-6. doi: 10.1016/j.jvn.2009.09.004. PMID 19914571
- [Background] Ho CK, Sun MP, Au TW, Chiu CS. Pneumatic pump reduces leg wound complications in cardiac patients. Asian Cardiovasc Thorac Ann. 2006 Dec;14(6):452-7. doi: 10.1177/021849230601400602. PMID 17130317
- [Background] Hassoun-Kheir N, Hasid I, Bozhko M, Shaban Z, Glam R, Hussein K, Paul M. Risk factors for limb surgical site infection following coronary artery bypass graft using open great saphenous vein harvesting: a retrospective cohort study. Interact Cardiovasc Thorac Surg. 2018 Oct 1;27(4):530-535. doi: 10.1093/icvts/ivy137. PMID 29688524
- [Background] Gulack BC, Kirkwood KA, Shi W, Smith PK, Alexander JH, Burks SG, Gelijns AC, Thourani VH, Bell D, Greenberg A, Goldfarb SD, Mayer ML, Bowdish ME; Cardiothoracic Surgical Trials Network (CTSN). Secondary surgical-site infection after coronary artery bypass grafting: A multi-institutional prospective cohort study. J Thorac Cardiovasc Surg. 2018 Apr;155(4):1555-1562.e1. doi: 10.1016/j.jtcvs.2017.10.078. Epub 2017 Dec 6. PMID 29221750
- [Background] Garland R, Frizelle FA, Dobbs BR, Singh H. A retrospective audit of long-term lower limb complications following leg vein harvesting for coronary artery bypass grafting. Eur J Cardiothorac Surg. 2003 Jun;23(6):950-5. doi: 10.1016/s1010-7940(03)00116-7. PMID 12829071
- [Background] Dusterhoft V, Bauer M, Buz S, Schaumann B, Hetzer R. Wound-healing disturbances after vein harvesting for CABG: a randomized trial to compare the minimally invasive direct vision and traditional approaches. Ann Thorac Surg. 2001 Dec;72(6):2038-43. doi: 10.1016/s0003-4975(01)03047-8. PMID 11789790
- [Background] Andrea Nelson E. Understanding compression therapy. J Wound Care. 1998 Jul 2;7(7):323. doi: 10.12968/jowc.1998.7.7.323. PMID 27966395
- [Background] Alizadeh-Ghavidel A, Ramezannejad P, Mirmesdagh Y, Sadeghpour-Tabaei A. Prevention of edema after coronary artery bypass graft surgery by compression stockings. Res Cardiovasc Med. 2014 May;3(2):e17463. doi: 10.5812/cardiovascmed.17463. Epub 2014 Apr 1. PMID 25478535
- See also: This study use the TED stockings after CABG and the protocol. such as the severity of edema and timing of follow up, from this study was used in my study. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4253792/
- See also: This study compare between stockings and conventional elastic bandages. The protocol, such as difference of circumference between preoperative leg and postoperative leg, was used in my study — https://pubmed.ncbi.nlm.nih.gov/19914571/
- See also: This paper proove that CPG-EB optimal subbandage pressure was not inferior than stockings. — https://pubmed.ncbi.nlm.nih.gov/27502619/

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-04-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT06603961/Prot_SAP_ICF_002.pdf